CLINICAL TRIAL: NCT04663269
Title: Randomized, Prospective Trial of Regional Erector Spinae Analgesic Block Versus Standard of Care in Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Regional Erector Spinae Analgesic Block vs Standard of Care Undergoing Percutaneous Nephrolithotomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Drop out from surgeons from 3 to 1. It will take too long to feasibly accrue with only one provider.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tim Large, Assistant Professor of Urology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 87943342
Record Dates: First submitted 2020-11-20; First posted 2020-12-10 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Kidney Stone; Surgery
MeSH Terms: conditions — Kidney Calculi | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Anesthesia will know the randomization assignment. The surgeon and the patient will be blinded to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Other): Standard Care Protocol - peritubal block standard local analgesic administration in the form of a peritubal block
  Interventions: Drug: Control Test
- ANES Block (Experimental): Patients randomized to the erector spinae block (Group 2) will have the block placed in the preoperative area by the anesthesia team. 0-4 mg midazolam and/or 0-100 mcg of fentanyl may be provided prior to and in order to place the block itself. The local anesthetic will diffuse to involve the dorsal and ventral rami of the spinal nerves, achieving a sensory block of the affected area. The erector spinae block analgesic will be administered by the anesthesia team. The analgesic provided in the erector spinae block is 20mL of 0.5% Bupivicaine with 4mg of PF Dexamethasone.
  Interventions: Drug: 4mg PF Dexamethasone

INTERVENTIONS:
Drug: 4mg PF Dexamethasone — analgesic provided in the erector spinae block is 20mL of 0.5% Bupivicaine with 4mg of PF Dexamethasone
  Arms: ANES Block
Drug: Control Test — Peritubal block - standard local analgesic administration
  Other Names: Standard of Care
  Arms: Control

SUMMARY:
The purpose of this study is to determine if adding a spinal block (medicine that will numb parts of the body to block pain) along with standard pain control at the incision site will decrease the need for narcotics for pain management and decrease the percentage of patients requiring hospital admission for pain control during postoperative , in-hospital, care after a percutaneous nephrolithotomy (PCNL) (surgery to remove kidney stones), commonly called PERC.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Undergoing unilateral or bilateral PCNL for treatment of kidney stones Estimated glomerular filtration rate > 30 mL/min. PCNL is planned as an outpatient procedure with no overnight hospital stay

Exclusion Criteria:

Inability to provide informed consent Pregnancy Patients having any additional simultaneous procedures other than a contralateral PCNL,(including contralateral treatment of kidney stones with a non-PCNL operation such as ureteroscopy) Patients with a documented neurologic injury that reduces pain sensation to the back Patients with an existing pain disorder Patients with an existing narcotics agreement due to current or prior narcotic abuse Patients with a documented allergy to a narcotic or NSAID analgesic BMI > 35 Patients who require more than 1 site of percutaneous access into the kidney to adequately complete the PCNL (this is a judgment made preoperatively at the initial clinic patient encounter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Overnight Admission Rate | 24 hours
  Percentage of patients in Groups 1 and 2 who require overnight admission to the hospital for pain control postoperatively (i.e. patients unable to be discharged to home from the postoperative anesthesia care unit PACU).

SECONDARY OUTCOMES:
Narcotic for Analgesia post-operatively | 14 days post-op
  Comparison of the percentage of patients in Groups 1 and 2 who require any narcotic for analgesia during the postoperative course following PCNL.
Proportion of patients with Emergency Department return or re-admission | 14 days
  Proportion of patient successfully discharged from PACU without return to Emergency Department or requiring re-admission within 14 days post discharge.
Number of Narcotic administrations post-operatively | 14 days
  Of patients requiring narcotics during the hospitalization, how many administrations of narcotics did these patients receive
Number of Morphine Equivalents post-operatively | 14 days
  Of patients requiring narcotics during the hospitalization, how many administrations of narcotics did these patients receive in daily morphine equivalents
Number of complications peri and post-operatively | 24 hours
  Any complications (according to Clavien-Dindo classification11) during the surgery and postoperative hospital stay
Pain Score | 24 hours
  Maximum patient reported pain score within the first 24 hours post operatively using 0-10 numeric pain intensity scale (NPIS) where 0 is no pain, 5 is moderate pain and 10 is the worst possible pain.
Rate of Adjunct Analgesics Post-operatively | 14 days
  Nonsteroidal Anti-inflammatories
  * Y/N
  * If Yes, name & dose
  * If Yes, total # of times administered
  * If Yes total # of times administered/(LOS in hours/24)
  Gabbapentinoids
  * Y/N
  * If Yes, name & dose
  * If Yes, total # of times administered
  * If Yes total # of times administered/(LOS in hours/24)
  Acetaminophen
  * Y/N
  * If Yes, name & dose
  * If Yes, total # of times administered
  * If Yes total # of times administered/(LOS in hours/24)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Large, MD, Principal Investigator — Indiana University
Locations (1):
- Methodist University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jonnavithula N, Pisapati MV, Durga P, Krishnamurthy V, Chilumu R, Reddy B. Efficacy of peritubal local anesthetic infiltration in alleviating postoperative pain in percutaneous nephrolithotomy. J Endourol. 2009 May;23(5):857-60. doi: 10.1089/end.2008.0634. PMID 19397429
- [Background] Parikh GP, Shah VR, Modi MP, Chauhan NC. The analgesic efficacy of peritubal infiltration of 0.25% bupivacaine in percutaneous nephrolithotomy - A prospective randomized study. J Anaesthesiol Clin Pharmacol. 2011 Oct;27(4):481-4. doi: 10.4103/0970-9185.86591. PMID 22096280
- [Background] Ozkan D, Akkaya T, Karakoyunlu N, Arik E, Ergil J, Koc Z, Gumus H, Ersoy H. Effect of ultrasound-guided intercostal nerve block on postoperative pain after percutaneous nephrolithotomy : prospective randomized controlled study. Anaesthesist. 2013 Dec;62(12):988-94. doi: 10.1007/s00101-013-2253-z. Epub 2013 Nov 1. PMID 24173546
- [Background] Honey RJ, Ghiculete D, Ray AA, Pace KT. A randomized, double-blinded, placebo-controlled trial of intercostal nerve block after percutaneous nephrolithotomy. J Endourol. 2013 Apr;27(4):415-9. doi: 10.1089/end.2012.0418. PMID 23445266
- [Background] Yang H, Yu X, Hu J, Peng E, Li C, Cui L, Zhao C, Wang S, Wei C, Mei W, Wang S, Ye Z. Usage of Multilevel Paravertebral Block as the Main Anesthesia for Mini-Invasive PCNL: Retrospective Review of 45 Cases with Large Stones. Urol Int. 2017;99(3):326-330. doi: 10.1159/000480094. Epub 2017 Aug 30. PMID 28850954
- [Background] Jonnavithula N, Chirra RR, Pasupuleti SL, Devraj R, Sriramoju V, Pisapati MV. A comparison of the efficacy of intercostal nerve block and peritubal infiltration of ropivacaine for post-operative analgesia following percutaneous nephrolithotomy: A prospective randomised double-blind study. Indian J Anaesth. 2017 Aug;61(8):655-660. doi: 10.4103/ija.IJA_88_17. PMID 28890561
- [Background] Hatipoglu Z, Gulec E, Turktan M, Izol V, Aridogan A, Gunes Y, Ozcengiz D. Comparative study of ultrasound-guided paravertebral block versus intravenous tramadol for postoperative pain control in percutaneous nephrolithotomy. BMC Anesthesiol. 2018 Feb 17;18(1):24. doi: 10.1186/s12871-018-0479-7. PMID 29454333
- [Background] Malekpour M, Hashmi A, Dove J, Torres D, Wild J. Analgesic Choice in Management of Rib Fractures: Paravertebral Block or Epidural Analgesia? Anesth Analg. 2017 Jun;124(6):1906-1911. doi: 10.1213/ANE.0000000000002113. PMID 28525509
- [Background] Yeying G, Liyong Y, Yuebo C, Yu Z, Guangao Y, Weihu M, Liujun Z. Thoracic paravertebral block versus intravenous patient-controlled analgesia for pain treatment in patients with multiple rib fractures. J Int Med Res. 2017 Dec;45(6):2085-2091. doi: 10.1177/0300060517710068. Epub 2017 Jun 21. PMID 28635359
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Miller NL, Matlaga BR, Lingeman JE. Techniques for fluoroscopic percutaneous renal access. J Urol. 2007 Jul;178(1):15-23. doi: 10.1016/j.juro.2007.03.014. Epub 2007 May 11. PMID 17574053